CLINICAL TRIAL: NCT06263101
Title: Drainage Fluid Biomarkers and Postoperative Gastrointestinal Dysfunction in Colorectal Surgery. A Monocentric Prospective Observational Study
Brief Title: Drainage Fluid Biomarkers and Postoperative Gastrointestinal Dysfunction in Laparoscopic Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Chaoyang Hospital of China Medical University (Other Government)
Responsible Party: Sponsor
Other Study IDs: ChaoyangHospital
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Gastrointestinal Dysfunction (POGD)
Keywords: postoperative ileus; drainage fluid; inflammatory markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Preoperative and postoperative blood samples. Postoperative drain fluid samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomarker-group: We considered for the study all patients diagnosed with colorectal cancer through preoperative colonoscopy, aged 18-80, underwent laparoscopic radical resection with confirmed pathology, without prior radiotherapy, chemotherapy, or immunotherapy, and voluntarily participated in and signed informed consent for the study, collected indicators of inflammation in the peripheral blood and post-operative drainage fluid of enrolled patients on post-operative days 1 and 3.
  Interventions: Other: Biochemical testing of abdominal drainage fluid; Other: Cytological examination of abdominal drainage fluid; Other: Peripheral blood cytology tests

INTERVENTIONS:
Other: Biochemical testing of abdominal drainage fluid — Drainage fluid was collected from patients on the first and third postoperative days to test the levels of three biochemical tests (albumin, lactate dehydrogenase [LDH], adenosine deaminase [ADA]).
Other: Cytological examination of abdominal drainage fluid — Cytological examination of abdominal drainage fluid on the first postoperative day and the third postoperative day, calculation of neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), prognostic nutritional index (PNI)
Other: Peripheral blood cytology tests — Peripheral blood cytology tests on the first postoperative day and the third postoperative day, calculation of Neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet lymphocyte ratio (PLR), systemic immunoinflammatory index (SII)

SUMMARY:
Postoperative gastrointestinal dysfunction (POGD), often referred to as postoperative ileus (POI) after colorectal surgery, is characterized by symptoms such as nausea, vomiting, abdominal distension, and delayed bowel movements. The incidence of this issue varies among medical institutions, impacting patient nutrition, prolonging hospital stays, and increasing healthcare costs.

The complex pathogenesis of POGD involves a brief neurogenic phase (within 3 hours) and a more prolonged inflammatory phase (beginning at 3-4 hours and lasting for days). The inflammatory phase is crucial and is recognized as initiated by mast cells and damage-associated molecular patterns that activate macrophages in the intestinal muscle layer. Subsequently, it triggers a series of cascading inflammation reactions through the release of inflammatory factors and recruitment of inflammatory cells, which contributes to the development and exacerbation of POGD. Studies have demonstrated changes in inflammatory cells and factors in the abdominal fluid following abdominal surgery, emphasizing the clinical significance of analyzing drainage fluid to predict postoperative gastrointestinal function.

This study analyzes inflammatory markers in drainage fluid following laparoscopic colorectal cancer surgery. The aim is to enhance the accuracy of predicting gastrointestinal recovery outcomes and contribute to the evolving field of Enhanced Recovery After Surgery (ERAS).

DETAILED DESCRIPTION:
Postoperative gastrointestinal dysfunction (POGD), often referred to as postoperative ileus (POI), is a common gastrointestinal issue that frequently occurs after colorectal surgery. It is characterized by symptoms such as nausea and vomiting, abdominal distension, and delayed defecation and evacuation. The incidence of POI is not clearly defined due to the varying definitions across healthcare institutions, but it is estimated to be approximately 10-30% and is one of the most common complications after colorectal surgery. The occurrence of POI increases the nutritional risk of patients (e.g., malnutrition, myasthenia gravis, malignant morbidity), prolongs the length of hospital stay, increases hospital costs, and significantly adds to the health economic burden.

In 2018, the American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement considered abandoning the traditional definition of POI and proposed a scoring system based on intake, sensation of nausea, vomiting, physical examination, and duration of symptoms (I-FEED). They also introduced a definition of postoperative gastrointestinal dysfunction (POGD) based on scores classifying postoperative gastrointestinal function as normal (0-2), postoperative gastrointestinal intolerance (POGI) (3-5), and postoperative gastrointestinal dysfunction (POGD) (>6).

The complex pathogenesis of POGD involves a brief neurogenic phase (within 3 hours) and a more prolonged inflammatory phase (beginning at 3-4 hours and lasting for days). The inflammatory phase is crucial and is recognized as initiated by mast cells and damage-associated molecular patterns that activate macrophages in the intestinal muscle layer. Subsequently, it triggers a series of cascading inflammation reactions through the release of inflammatory factors and recruitment of inflammatory cells, which contributes to the development and exacerbation of POGD.

Levels of inflammatory cells and factors in the peritoneal fluid are changed following abdominal surgery in both rodents and humans. Many previous studies have confirmed that the use of drainage fluids also reduces the incidence of elevated inflammatory markers, such as CRP, in the presence of unrelated inflammatory stimuli, such as concurrent infections and systemic diseases. For instance, in other diseases like meningitis, blood IL-6 is less specific than IL-6 in the drainage fluid. In addition, abdominal drainage fluid is more effective and efficient than routinely collected blood for detecting anastomotic leakage (AL) following colorectal cancer surgery. However, fewer studies have been conducted to predict the recovery of postoperative gastrointestinal function by analyzing drainage fluid. We believe that analyzing postoperative gastrointestinal drainage fluid is of greater clinical importance in predicting postoperative gastrointestinal function.

In our study, we collected abdominal drainage fluid near the anastomosis on the first and third day after laparoscopic colorectal cancer surgery for biochemical and cytological tests. These tests included lactate dehydrogenase (LDH), adenosine deaminase (ADA) and albumin. We also performed conventional cytological tests for neutrophils, lymphocytes, monocytes, etc. In addition, we calculated inflammatory indices such as neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR) and prognostic nutrition index (PNI). We also collected peripheral blood for the same cytological indices and evaluated the outcome of the patients' gastrointestinal function recovery using the I-FEED score. In addition, we analyzed the correlation between the above indices and PODG, and combined the inflammation indices of peritoneal drainage and serum to predict the outcome of gastrointestinal function recovery after laparoscopic colorectal cancer surgery aiming to improve the accuracy and effectiveness of prediction and accelerate patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative diagnosis of colorectal cancer through colonoscopy biopsy.
* Patients aged 18-80 years.
* Underwent laparoscopic radical resection for colorectal cancer with confirmed postoperative pathology.
* No prior radiotherapy, chemotherapy, or immunotherapy before surgery.
* Voluntary participation in the study and signing of a written informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* Severe liver dysfunction (Child-Pugh class B or above); severe renal dysfunction (serum creatinine level greater than 177).
* Patients with severe heart failure, chronic obstructive pulmonary disease, and other underlying diseases.
* Patients with pre-existing severe infections (developing sepsis or not improving after antibiotic treatment) before surgery.
* Patients with postoperative fistulas or those requiring a two-stage anastomosis.
* Intraoperative and postoperative intraperitoneal chemotherapy.
* Blood disorders (leukemia, lymphoma, aplastic anemia, etc.).
* Patient or family member withdraws midway.
* Those with serious post-operative infections (e.g., incisional, lung, and urinary tract infections)
* Intraoperative conversion to open laparotomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 with preoperative colorectal cancer diagnosis through colonoscopy biopsy underwent laparoscopic radical resection, excluding prior radiotherapy, chemotherapy, or immunotherapy, and voluntarily participated by signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Measurement of drainage fluid LDH and neutrophil to lymphocyte ratio (NLR) on postoperative day 1 | Postoperative day 1
  Our primary endpoint was to assess the role of drainage fluid LDH and neutrophil to lymphocyte ratio (NLR) on postoperative day 1.

SECONDARY OUTCOMES:
Measurement of drainage fluid LDH and neutrophil to lymphocyte ratio (NLR) on postoperative day 3 | Postoperative day 3
  Our Secondary endpoint was to assess the role of drainage fluid LDH and neutrophil to lymphocyte ratio (NLR) on postoperative day 3.
Measurement of drainage fluid albumin, adenosine deaminase (ADA), a d lymphocyte-monocyte ratio (LMR) on postoperative day 1 | Postoperative day 1
  Our Secondary endpoint was to assess the role of drainage fluid albumin, adenosine deaminase (ADA),and lymphocyte-monocyte ratio (LMR) on postoperative day 1.
Measurement of drainage fluid albumin, adenosine deaminase (ADA), lymphocyte-monocyte ratio (LMR) on postoperative day 3 | Postoperative day 3
  Our Secondary endpoint was to assess the role of drainage fluid albumin, adenosine deaminase (ADA),and lymphocyte-monocyte ratio (LMR) on postoperative day 3.
Measurement of blood serum neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet-lymphocyte ratio (PLR), systemic immune-inflammatory index (SII) on postoperative day 1. | Postoperative day 1
  Our Secondary endpoint was to assess the role of blood serum neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet-lymphocyte ratio (PLR), systemic immune-inflammatory index (SII) on postoperative day 1.
Measurement of blood serum neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet-lymphocyte ratio (PLR), systemic immune-inflammatory index (SII) on postoperative day 3. | Postoperative day 3
  Our Secondary endpoint was to assess the role of blood serum neutrophil-lymphocyte ratio (NLR), lymphocyte-monocyte ratio (LMR), platelet-lymphocyte ratio (PLR), systemic immune-inflammatory index (SII) on postoperative day 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaoyang Central Hospital of China Medical University, Chaoyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chapman SJ, Pericleous A, Downey C, Jayne DG. Postoperative ileus following major colorectal surgery. Br J Surg. 2018 Jun;105(7):797-810. doi: 10.1002/bjs.10781. Epub 2018 Feb 22. PMID 29469195
- [Background] Scarborough JE, Schumacher J, Kent KC, Heise CP, Greenberg CC. Associations of Specific Postoperative Complications With Outcomes After Elective Colon Resection: A Procedure-Targeted Approach Toward Surgical Quality Improvement. JAMA Surg. 2017 Feb 15;152(2):e164681. doi: 10.1001/jamasurg.2016.4681. Epub 2017 Feb 15. PMID 27926773
- [Background] Iyer S, Saunders WB, Stemkowski S. Economic burden of postoperative ileus associated with colectomy in the United States. J Manag Care Pharm. 2009 Jul-Aug;15(6):485-94. doi: 10.18553/jmcp.2009.15.6.485. PMID 19610681
- [Background] Hedrick TL, McEvoy MD, Mythen MMG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Postoperative Gastrointestinal Dysfunction Within an Enhanced Recovery Pathway for Elective Colorectal Surgery. Anesth Analg. 2018 Jun;126(6):1896-1907. doi: 10.1213/ANE.0000000000002742. PMID 29293183
- [Background] Wehner S, Behrendt FF, Lyutenski BN, Lysson M, Bauer AJ, Hirner A, Kalff JC. Inhibition of macrophage function prevents intestinal inflammation and postoperative ileus in rodents. Gut. 2007 Feb;56(2):176-85. doi: 10.1136/gut.2005.089615. Epub 2006 Jun 29. PMID 16809419
- [Background] Bauer AJ. Mentation on the immunological modulation of gastrointestinal motility. Neurogastroenterol Motil. 2008 May;20 Suppl 1:81-90. doi: 10.1111/j.1365-2982.2008.01105.x. PMID 18402645

DOCUMENTS (3):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06263101/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06263101/SAP_001.pdf
  • Informed Consent Form (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06263101/ICF_002.pdf